CLINICAL TRIAL: NCT04421326
Title: Multimodal Investigation of Intracranial Clot Environment
Acronym: MISO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Genomic Institute of Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0236
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Acute Ichemic Stroke; Brain Ischemia
Keywords: Stroke; Blood Brain Barrier; Ischemia; Thrombus; Interventional Neuroradiology
MeSH Terms: conditions — Brain Ischemia; Stroke; Ischemia; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute ischemic stroke: Patients undergoing Mechanical Thrombectomy for large vessel occclusion with acute ischemic stroke
  Interventions: Other: Analysis of the clot

INTERVENTIONS:
Other: Analysis of the clot — Blood sampling at the site of intracranial occlusion during Mechanical Thrombectomy

SUMMARY:
Analysis of peri clot blood collected at the acute phase of stroke in order to understand physiopathological mechanisms involved in the cerebrovascular damage

DETAILED DESCRIPTION:
It has been shown that immune cells accumulate around the clot at the acute phase of stroke. Leukocytes and their specific chemokines and cytokines regulation may impact cerebrovascular integrity.

ELIGIBILITY:
Inclusion criteria:

1. Over 18 years of age,
2. Non-dependent for activities of daily living prior to the onset of the MI (Modified Rankin Score >2)
3. Having an occlusion of a large arterial trunk proven by imaging (angio-MRI or angio-scanner).

Exclusion criteria:

1. Patients initially admitted but for whom endovascular treatment will not finally be performed (re-infusion, catheterization failure...) will be excluded from the study.
2. Major patients under guardianship or curatorship or patients deprived of liberty

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Mechanical Thrombectomy for large vessel occclusion with acute ischemic stroke
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Metalloproteinase 9 quantification | 60 months
Metalloproteinase 2 quantification | 60 months

SECONDARY OUTCOMES:
Cytokines levels | 60 months
  Proteomic analysis of cytokines IL-1β, TNF-α, IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Vincent COSTALAT, MD PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No